CLINICAL TRIAL: NCT05362370
Title: Stryker PEEK Customized Implant: A Prospective Post Market Follow Up to Evaluate Safety, Performance and Effectiveness
Status: Recruiting | Type: Observational
Sponsor: Stryker Craniomaxillofacial (Industry)
Collaborators: Qmed Consulting A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CMF_2021_01
Record Dates: First submitted 2022-04-12; First posted 2022-05-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cranioplasty; Craniofacial Abnormalities; Craniofacial Injuries
MeSH Terms: conditions — Craniofacial Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Participants will receive a Stryker PEEK Customized Implant
  Interventions: Device: Stryker's PEEK Customized Implant

INTERVENTIONS:
Device: Stryker's PEEK Customized Implant — The PEEK Customized Implants will be used in this patient cohort for augmentation and/or restoration of bony and/or soft tissue deformities in the cranial and craniofacial skeleton (orbital rim, zygoma, and adjacent bone); including but not limited to, the correction and prevention of persistent temporal hollowing (PTH).

SUMMARY:
The purpose of this study is to confirm the safety, performance and effectiveness of Stryker's PEEK Customized Implants when used for the augmentation and/or restoration of bony and/or soft tissue deformities in the cranial and craniofacial skeleton. The study is designed as a prospective, multi-center trial with a long-term follow-up (24 months) of study participants.

DETAILED DESCRIPTION:
Stryker's PEEK Customized Implants are patient-specific implants based on CT-data of the individual patient and input of the surgeon. The implants are fabricated from Polyetheretherketone (PEEK) and intended to be used to fill bony voids in the cranial and craniofacial region (e.g. cranium, orbital rim, zygoma, and adjacent bone). This observational post-market clinical follow-up (PMCF) is designed to confirm the safety, performance and clinical benefit of Stryker's PEEK Customized Implants for the augmentation and/or restoration of bony and/or soft tissue deformities in the cranial and craniofacial skeleton (orbital rim, zygoma, and adjacent bone); including but not limited to, the correction and prevention of persistent temporal hollowing (PTH). Infection of implants is one of the common risks associated with this type of surgery. This PMCF study will investigate infection rate as the primary safety endpoint. These data will be collected in a real world setting, where all treatment is per routine clinical practice. The study is designed as a prospective, multi-center trial at participating institutions in the United States and in Europe. Up to 110 study participants will be enrolled in this PMCF. Stryker's PEEK Customized Implants are intended to stay implanted permanently. Therefore, study participants will be followed for 24 months after implantation of the devices to allow evaluation of long-term safety and performance of the products.

ELIGIBILITY:
Inclusion Criteria

1. Subject is eligible for a PEEK customized implant as per routine clinical practice.
2. Subject is 12 years of age or older (Europe only).
3. Subject is 3.5 years of age or older (USA only).
4. Adult subjects able to give consent.
5. Subjects under the age of 18 will have a legal representative or parents (France - both parents must sign) to provide informed consent.
6. Subjects who are unable to give consent themselves but have a legally authorized representative that may consent on their behalf.

Exclusion Criteria

1. Subject has an active systemic or local infection.
2. Subject has known allergy to plastic or polymers and/or known sensitivity to foreign bodies.
3. Comprised bone due to poor blood supply, disease, infection or prior implantation, which would not allow adequate support or fixation of the implant.
4. Mental or neuromuscular disorder which could create an unacceptable risk of implant instability or implant fixation failure, or complications in postoperative care.
5. Knowingly pregnant or nursing women.
6. Concomitant participation in other clinical trials related to cranioplasty.
7. Subject who has an expected survival rate of less than 2 years, in the opinion of the investigator who takes consent.

Min Age: 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cranial and craniofacial defects requiring augmentation and/or restoration, e.g. following tumor resection, trauma, vascular conditions, or stroke requiring craniectomy, due to previously failed cranioplasty, or bone flap resorption.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Infection Rate | 24 months post-operative
  Assessment of rate of infection associated with Stryker's PEEK Customized Implants.

SECONDARY OUTCOMES:
Incidence of device related serious adverse events (SAEs) | 24 months post-operative
  Incidence of device related SAEs up to 24 months post implantation
Ability to place the Customized Implant during surgery leading to good aesthetic outcome | 24 months post-operative
  Assessment of success of placement by the surgeon as determined by the ability to close the defect effectively, even with modification of implant
Rate of implant failure | 24 months post-operative
  Rate of implant failure leading to explantation
Quality of life questionnaire | 24 months post-operative
  Outcome of Short Form health survey-12 (SF-12) quality of life questionnaire
Length of hospitalisation | Up to 1 month
  Time duration after surgery until hospital discharge
Persistent temporal hollowing | 24 months post-operative
  Presence of persistent temporal hollowing after the procedure
Neurological Assessment | 24 months post-operative
  Glasgow Coma Scale
Scale of brain injuries | 24 months post-operative
  Glasgow Outcome Scale Extended
Aesthetic assessment | 24 months post-operative
  Aesthetic assessment score

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - University of Louisville 501 E. Broadway, Suite 210, Louisville, Kentucky
  - Department of Neurological Surgery, New Brunswick, New Jersey
  - Department of Neurological Surgery, 710 West 168th Street, 4th Floor, New York Presbyterian Hospital, New York, New York
  - Lewis Katz School of Medicine at Temple University, 3401 North Broad Street, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Oral & Maxillofacial Surgery, 173 Ashley Avenue, Charleston, USA, Charleston, South Carolina
- Universitätsklinik für Neurochirurgie Auenbruggerplatz 29, Graz, Austria
- France (3):
  - Pierre-Paul Riquet Hospital, Place du Docteur Baylac, Cedex 9, Toulouse, Occitanie
  - APHP - Hôpital Lariboisière Neurochirurgie 2 rue Ambroise Paré, Paris, Paris France
  - CHU Nantes - Hopital Guillaume et Rene Laënnec, Cedex 1, Nantes, Pays de la Loire Region
- Germany (2):
  - St. Barbara-Klinik Hamm GmbH Hamm Heessen und St. Josef-Krankenhaus Hamm-Bockum-Hövel Am Heessener Wald 1 | 1263, Hamm, Hamm
  - Klinik für Neurochirurgie Klinikum Dortmund Münsterstr. 240, Dortmund, North Rhine-Westphalia
- Servicio de Neurocirugía Hospital Universitario La Paz., Madrid, Madrid, Spain
- Neurosurgery, Emergency and Major Trauma (NET) Research | Division of Medicine | Imperial College Healthcare NHS Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No